CLINICAL TRIAL: NCT03343964
Title: Can Bedside Amplitude-integrated EEG Improve Seizure Detection and Prognostication in Children With Traumatic Brain Injury in a Hospital With Limited Access to Conventional EEG?
Brief Title: Amplitude-integrated EEG in Improvement of Seizure Detection and Prognostication in Children With TBI
Acronym: aEEG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Genevieve Du Pont-Thibodeau (Other)
Responsible Party: Sponsor-Investigator, Genevieve Du Pont-Thibodeau, Pediatric intensivist, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Other Study IDs: CHUSJ 2018-1556
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Traumatic Brain Injury
Keywords: aEEG, cEEG
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with moderate to severe TBI
  Interventions: Diagnostic Test: Amplitude-integrated electroencephalography

INTERVENTIONS:
Diagnostic Test: Amplitude-integrated electroencephalography — Amplitude-integrated EEG (aEEG) is a compressed form of real-time conventional EEG monitoring that will be added to cEEG monitoring.

SUMMARY:
The goal of this study is to determine whether the addition of aEEG to cEEG in clinical practice does in fact help PICU physicians detect subclinical seizures in this population.

DETAILED DESCRIPTION:
Children with moderate to severe TBI are at risk of significant long-term neurological sequelae. Careful post-injury management is crucial in optimizing their recovery. Seizures are a frequent complication. They are associated with worse outcome and require prompt intervention. However, they are often subclinical and are only detectable by gold-standard conventional electroencephalography (cEEG); a costly, complex monitoring device that is not readily available 24/7 in many pediatric intensive care units (PICUs) and can only be interpreted by neurologists. On average, PICUs obtain only 1-2 cEEG reports per day from neurologists and this can lead to significant delays in seizure identification and treatment. Amplitude-integrated EEG (aEEG) is a compressed form of real-time cEEG monitoring that can be added to cEEG monitoring. It is more easy to interpret and can be taught to PICU providers with limited training. It is a promising complementary tool that could help PICU physicians identify subclinical seizures and treat seizures more promptly. This could significantly improve the global outcome of this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe TBI defined by a post-resuscitation Glasgow Coma Scale (GCS) of 3-8 (severe) or 9-12 (moderate), this includes those with accidental TBI, abusive head trauma, and cases of polytrauma
* decision by the primary medical team to initiate cEEG monitoring

Exclusion Criteria:

* patients for whom it is impossible to record cEEG for any reason will be excluded from the study
* premature neonates
* brain death or suspected brain death at PICU entry
* unavailable equipment for cEGG and/or aEEG
* consent to participate denied by parents and/or patient

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients admitted to the Pediatric Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
accuracy of PICU physicians at detecting seizures when using aEEG in real-life clinical setting during the continuous EEG monitoring of patients with moderate to severe TBI | 18 months
  PICU physicians should correctly detect > 70% of all subclinical seizures. False positives rates should be < 20%.

SECONDARY OUTCOMES:
Determine whether a 2-hour aEEG teaching session is sufficient for PICU physicians to achieve similar seizure detection rates as experts in aEEG interpretation. | 18 months
  After a 2 hour aEEG training session, PICU physicians should have similar sensitivity and false positive rates as experts in aEEG.
Determine whether aEEG background activity correlates with patients' neurological outcome. | 18 months
  Continuous and reactive backgrounds should correlate with a good neurological outcome. Low voltage, discontinuous or burst suppression backgrounds should correlate with a poor neurological outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Du Pont-Thibodeau, MD, MSc, Principal Investigator — Sainte-Justine University Hospital Research Centre
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No